CLINICAL TRIAL: NCT00232323
Title: Experimental Like Study of Stress Reduction in Intensive Care Teams by Use of Simulation Training
Brief Title: Simulation Training as a Tool to Decrease Occupational Stress in ICU Personnel
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: SHEBA-05-3711-AN-CTIL
Record Dates: First submitted 2005-10-02; First posted 2005-10-04 (Estimated); Last update posted 2007-01-24 (Estimated); Status verified 2007-01

CONDITIONS: Education, Health
Keywords: intensive care; stress; education; simulation
MeSH Terms: conditions — Health Education

INTERVENTIONS:
Behavioral: simulation training

SUMMARY:
The purpose of the study is to check wether training mixed teams of physicians and nurses from intensive care units on patient simulators reduces stress in team members.

DETAILED DESCRIPTION:
Patient safety and the prevention of medical error are primary goals of healthcare organizations. Stress reduction may reduce or ameliorate such errors. Simulation training, using advanced patient simulators, has been shown to improve diagnostic, resuscitation and technical skills amongst physicians and nurses.We intend to check wether stress during ICU shifts may be reduced by using specifically designed scenarios based on real life experience,in integrative multidisciplinary ICU teams.

ELIGIBILITY:
Inclusion Criteria:

* intensive care physicians and nurses working in respiratory ICU willing to participate in the study

Exclusion Criteria:

* unwilling to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2006-01; Study Completion 2006-06

PRIMARY OUTCOMES:
reduction of stress parameters

CONTACTS AND LOCATIONS:
Overall Officials: Asaph E Nini, MD, Principal Investigator — Sheba Medical Center and Medical Simulation Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel